CLINICAL TRIAL: NCT05540002
Title: Efficacy of the Quell Wearable Device for Treatment of Central Sensitization-related Pain Among Persons With Chronic Overlapping Pain Conditions
Brief Title: Efficacy of the Quell Wearable Device for Chronic Overlapping Pain Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Robert N. Jamison, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P002083
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Adults 21 and Older; Multiple Chronic Overlapping Pain Conditions; Hypersensitivity
Keywords: Multiple Chronic Overlapping Pain Conditions; Adults 21 and older
MeSH Terms: conditions — Chronic Pain; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Participants will be equally randomized to one of the two treatment groups: the High Intensity Quell group or the Low Intensity Quell group. All groups will receive the same questionnaires and undergo quantitative sensory testing.
Who Masked: Participant, Investigator
Masking Description: Neither the principal investigator, the co-investigators, the research assistant, or the subjects will know if they are given the high intensity Quell device or the low intensity Quell device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High Intensity Stimulation (Active Comparator): Patients will be randomly assigned to the High Intensity Quell group and will receive higher intensity stimulation every day for 12 weeks.
  Interventions: Device: High Intensity Quell
- Low Intensity Stimulation (Sham Comparator): Patients will be randomly assigned to the Low intensity Quell group and will receive lower intensity stimulation every day for 12 weeks.
  Interventions: Device: Low Intensity Quell

INTERVENTIONS:
Device: High Intensity Quell — Participants will receive 1 hour of continuous stimulation during each therapy session. Subjects are asked to complete a minimum of 3 sessions per day.
  Arms: High Intensity Stimulation
Device: Low Intensity Quell — Participants will receive only three 2-minute periods of stimulation (at 0, 28, 58 minutes) during each 60-minute therapeutic session. Subjects are asked to complete a minimum of 3 sessions per day.
  Arms: Low Intensity Stimulation

SUMMARY:
This study will examine the pain-relieving effects of a transcutaneous electrical nerve stimulator device called a Quell for persons with multiple chronic overlapping pain conditions.

DETAILED DESCRIPTION:
This study will examine the pain-relieving effects of a transcutaneous electrical nerve stimulator device called a Quell for persons with multiple chronic overlapping pain conditions. Participants will attend two quantitative sensory testing visits in order to determine their level of pain sensitivity, one at the beginning of the study and the second at the 3-month Follow-up session. Participants will be asked to test out the Quell device to check for sensation tolerance, and will then be randomized into one of the two treatment groups: the High Intensity Quell group or the Low Intensity Quell group. Participants will be asked to wear the device for at least 3 hours every day and to complete daily assessments, along with a total of three sets of questionnaires: one at the start of the study, the second 6 weeks from the date of consent, and the third 3 months after the date of consent. A member of the research staff will call participants once a week for a brief phone interview throughout the study. Participants will be in this study for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 and older
* Pain duration > 3 months
* Diagnosed by physician with multiple chronic pain conditions
* Have chronic pain related to multiple chronic pain diagnoses (headaches, joint pain, back pain, or any of the other COPCs)
* Average 4 or greater on pain intensity scale of 0 to 10
* Pain is not accounted for by any other progressive disease (e.g., cancer, MS)
* Meets sensory hypersensitivity cutoffs based on QST-assessed evidence
* Own a smartphone (iPhone or Android device) and can download the pain app (MasterMyPain) and the Quell Relief mobile app onto their device
* Able to speak and understand English

Exclusion Criteria:

* Diagnosis of cancer or any other malignant disease
* Acute osteomyelitis or acute bone disease
* Present of past DSM-V diagnosis of schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder that would be judged to interfere with study participation
* Pregnancy
* Any clinically unstable systemic illness judged to interfere with treatment
* A pain condition requiring urgent surgery
* An active substance use disorder, such as cocaine or IV heroin use that would interfere with study participation
* Have an implanted cardiac pacemaker, defibrillator, or other implanted device.
* Reynaud's syndrome
* Open cuts/sores

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Jamison, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital Pain Management Center, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to rally website to Quell COPCs — http://rally.massgeneralbrigham.org/study/_quellcopcs

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Started | 58 | 57
Completed | 52 | 50
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 41 | 87
  >=65 years | 12 | 16 | 28
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 5 | 12 | 17
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 52 | 49 | 101
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 43 | 44 | 87
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Brief Pain Inventory Interference Scale (BPI)
Description: This is a validated measure of combined activity interference on a numerical scale of 0-10, with higher scores representing greater activity interference. We collected ratings on how much pain interfered over the past 24 hours with 1) General activity, 2) Mood, 3) Walking ability, 4) Normal work, 5) Relations with other people, 6) Sleep, and 7) Enjoyment of life on a scale of 0=does not interfere to 10=completely interferes. The table represents combined mean scores between groups. These ratings were collected at 3 months after start of the study.
Time Frame: Between group differences at 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 5.7 (1.7) | 5.7 (2.2)

2. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: Measures thoughts and feelings when patient is experiencing pain on a 13-item scale ranging from 0-52 with higher scores meaning a worse outcome and higher catastrophizing
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 25.0 (11.6) | 24.8 (13.3)

3. Secondary Outcome: Pain Disability Index (PDI)
Description: Rating scales designed to measure levels of pain disability, or the degree to which pain is preventing a patient from doing what they normally would be doing, or doing it as well as they normally would on a 7-item scale of 0-10 ranging from 0-70 with higher scores meaning a worse outcome
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 38.3 (14.6) | 36.3 (16.8)

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Measures mood on a 14-item scale ranging from 0 to 42 with higher scores meaning a worse outcome
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 19.1 (7.7) | 16.9 (7.8)

5. Secondary Outcome: Pain Detect Neuropathic Pain Questionnaire (painDETECT)
Description: Measures the presence of neuropathic pain on a scale ranging from 1 to 38 on ratings of 'never to very strongly' with higher scores meaning a worse outcome
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 16.1 (7.6) | 16.5 (7.4)

6. Secondary Outcome: Symptom Impact Questionnaire (SIQR)
Description: Measures 20 pain symptoms and function on a scale of 0-10 with scores ranging from 0 to 200 with higher scores meaning a worse outcome
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 115.8 (37.4) | 106.1 (38.9)

7. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: Measures the subject's overall belief about the efficacy of treatment on a 7-point categorical verbal rating scale. The scale ranges from (1) "no change or condition has gotten worse" to (7) "a great deal better and a considerable improvement that has made all the difference.
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 4.2 (1.8) | 4.0 (2.0)

8. Secondary Outcome: Healthcare Utilization
Description: Monthly clinic and ED visits
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
Number of visits
  Clinic visits | 1.3 (1.1) | 1.6 (1.7)
  Hospital visits | 0.0 (0.2) | 0.1 (0.2)

9. Secondary Outcome: Satisfaction and Qualitative Questions
Description: A satisfaction questionnaire was developed for this study specifically related to use of the pain management device (Quell) and use of the study app. Ten items related to use of the device and five items were related to use of the smartphone study app all rated on a scale of 0 (worse) to 10 (better). Below are group differences on "How willing would you be to using the Quell in the future?" rated from 0=Not at all willing to 10=Very willing. This questionnaire was only administered at the end of the trial.
Time Frame: 3-month Follow-up
Measure: Mean (Standard Deviation); unit: score on a 0-10 scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a 0-10 scale | 7.6 (2.9) | 7.4 (2.7)

10. Secondary Outcome: Quantitative Sensory Testing (QST)
Description: Set of psychophysical methods used to quantify somatosensory function. Combined hypersensitivity measure that measures responses to repeated touch, mechanical/pressure pain assessment, and cold pain assessment. Overall sensitivity based on z scores categorized into high and low sensitivity. Higher scores represent less sensitivity. The mean score is 0.
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 0.6 (2.0) | 0.0 (2.0)

11. Secondary Outcome: The Brief Pain Inventory Pain Intensity Scale (BPI)
Description: Average pain on a scale of 0-10 with higher scores meaning a worse outcome
Time Frame: Changes from Baseline to 3-month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | -0.5 (2.5) | -1.0 (2.3)

12. Secondary Outcome: MasterMyPain App
Description: Daily ratings of pain related factors on smartphone pain app on a scale of 0-10 with higher scores meaning a worse outcome. Multiple daily assessments were averaged for mean and standard deviation scores.
Time Frame: Daily ratings over 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
Number analyzed (Participants) | 58 | 57
score on a scale | 3.9 (3.2) | 5.1 (3.3)

ADVERSE EVENTS:
Time Frame: During the 3-month trial
Arm/Group | High Intensity Stimulation | Low Intensity Stimulation
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 19/58 | 14/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Intensity Stimulation (N=58) | Low Intensity Stimulation (N=57)
Related (General disorders) | 9 | 6
Unrelated (General disorders) | 10 | 8

LIMITATIONS AND CAVEATS:
There were several limitations. The study included a limited number of subjects. Subjects were only followed for 3 months. The subjects had other medical comorbidities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT05540002/Prot_SAP_000.pdf